CLINICAL TRIAL: NCT01563913
Title: Reducing Dyskinesia in Parkinson Disease With Omega-3 Fatty Acids
Brief Title: Reducing Dyskinesia in Parkinson's Disease With Omega-3 Fatty Acids
Acronym: RLID-PD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CLIN-006-11S; 2907 (Other: Portland VA Medical Center); 8012 (Other: Oregon Health & Science University)
Record Dates: First submitted 2012-03-16; First posted 2012-03-27 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinsons disease; supplement; DHA; dyskinesia; abnormal movements
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Docosahexaenoic Acids; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Docosahexaenoic Acid (DHA)
  Interventions: Drug: Docosahexaenoic Acid (DHA)
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Docosahexaenoic Acid (DHA) — Docosahexaenoic Acid (DHA) 2 grams per day taken for 1.5 years
  Other Names: DHA
  Arms: Arm 1
Drug: Placebo — Sugar Pill, taken for 1.5 years
  Other Names: Sugar Pill
  Arms: Arm 2

SUMMARY:
The purpose of this research study is to measure the safety (side effects) of an Omega 3 Fatty acid called docosahexanoic acid (DHA) and measure the dyskinesia (involuntary movements) in Parkinson 's disease (PD).

DETAILED DESCRIPTION:
Levodopa induced dyskinesias (LID) are involuntary, abnormal movements that occur in most patients with Parkinson disease(PD) as a consequence of chronic use of the most effective symptomatic drug, levodopa (LD). LID can range from subtle and unobtrusive to marked and disabling. There are surprisingly few treatments for LID, including amantadine and deep brain stimulation. In many instances, amantadine is either poorly tolerated, or provides inadequate benefit, and only a small minority are appropriate candidates for surgery. Given the finding that docosahexanoic acid (the most abundant omega-3 fatty acid in the brain), delays the onset and reduces the severity of dyskinesia in two different animal models of LID, a trial of docosahexanoic acid (DHA) in PD subjects about to start LD as part of their drug regimen, to prevent or slow the progression of LID is warranted.

Prior to embarking on a large trial, preliminary data about safety and tolerability of DHA in PD subjects is needed, and collection of this data is the primary outcome of this pilot project proposal. 40 subjects who have not yet used levodopa, but are about to begin it will be randomized to daily DHA or placebo. Safety laboratory testing, adverse event monitoring, DHA plasma and CSF levels as well as compliance/subject retention will be outcomes collected.

In addition, preliminary data about modification of incidence rates will be collected and compared between the two treatment groups. This information will aid in calculating an appropriate sample size and treatment period for a larger definitive future study.

Dyskinesia manifests overwhelmingly when plasma levodopa levels are high enough to cause anti-parkinsonian benefits, and lessens or stops when levodopa levels drop below a threshold. Thus, the subject's dyskinesia measurements must occur during a levodopa administration period. Dyskinesia measurement will occur during a two-hour levodopa cycle administered to subjects at weeks 0, 6, 24, 52, 76. It is expected that a good proportion of subjects will manifest dyskinesia within the two-year observation period, as previous studies using the most objective means to measure dyskinesia report incidence rates of 67% or greater within the first year of levodopa use. An instrument to measure dyskinesia developed by this center will be used as an additional outcome, and is expected to measure dyskinesia more accurately and with greater sensitivity than the gold standard methods of clinical rating scales.

By conclusion of this pilot project, the safety and tolerability, subject retention and compliance, plasma/CSF levels of DHA administration will be determined. Trends in dyskinesia development may be measured. This will provide the needed background information to proceed with a future larger trial of DHA to prevent dyskinesia in PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinsons disease
* No levodopa (Sinemet) treatment or prior exposure to levodopa

Exclusion Criteria:

* Prior exposure to levodopa
* Unable to stand for 1 minute without aid
* Sensory deficits on feet
* Significant cognitive impairment
* Current use of dopamine receptor blocking medications (depakote, lithium, amiodarone, tetrabenazine, metoclopramide, dronabinol)
* Current fish oil or lutein supplementation
* Allergy to soy

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Anne Chung, MD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salem N Jr, Litman B, Kim HY, Gawrisch K. Mechanisms of action of docosahexaenoic acid in the nervous system. Lipids. 2001 Sep;36(9):945-59. doi: 10.1007/s11745-001-0805-6. PMID 11724467
- [Result] Pechevis M, Clarke CE, Vieregge P, Khoshnood B, Deschaseaux-Voinet C, Berdeaux G, Ziegler M; Trial Study Group. Effects of dyskinesias in Parkinson's disease on quality of life and health-related costs: a prospective European study. Eur J Neurol. 2005 Dec;12(12):956-63. doi: 10.1111/j.1468-1331.2005.01096.x. PMID 16324089
- [Result] Rascol O, Brooks DJ, Korczyn AD, De Deyn PP, Clarke CE, Lang AE. A five-year study of the incidence of dyskinesia in patients with early Parkinson's disease who were treated with ropinirole or levodopa. N Engl J Med. 2000 May 18;342(20):1484-91. doi: 10.1056/NEJM200005183422004. PMID 10816186
- [Result] Nutt JG, Carter JH, Lea ES, Sexton GJ. Evolution of the response to levodopa during the first 4 years of therapy. Ann Neurol. 2002 Jun;51(6):686-93. doi: 10.1002/ana.10189. PMID 12112073
- [Result] Chung KA, Lobb BM, Nutt JG, McNames J, Horak F. Objective measurement of dyskinesia in Parkinson's disease using a force plate. Mov Disord. 2010 Apr 15;25(5):602-8. doi: 10.1002/mds.22856. PMID 20213818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from two large urban hospitals with Movement disorder specialty clinics in the NW USA over a 30 month (2.5 year) recruitment period. 34 subjects were screened. 1 subject screen failed due to prior exposure to levodopa. 33 subjects were randomized to DHA or placebo arms. 30 subjects returned and completed visit 1.
Period: Overall Study
Arm/Group | Docosahexaenoic Acid (DHA) | Placebo
Started | 15 | 15
Completed | 13 | 15
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Spouse Passed Away | 1 | 0

BASELINE CHARACTERISTICS:
Population: Report on the participants that were randomized and completed visit 1.
Groups:
- Docosahexaenoic Acid: Docosahexaenoic Acid (DHA) 2 grams per day taken for 1.5 years
- Placebo:: Placebo: Sugar Pill, taken for 1.5 years
- Total: Total of all reporting groups
Arm/Group | Docosahexaenoic Acid | Placebo: | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (7.6) | 67.0 (8.5) | 68.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Large Northwest American City
  Participants
    United States | 15 | 15 | 30
PD Symptom Duration [Mean (Standard Deviation); unit: years] — Year of screening visit - Subjectively reported onset of Parkinson's symptoms year
  years | 3.2 (1.9) | 4.6 (3.8) | 3.8 (2.9)
Education [Mean (Standard Deviation); unit: years] — Number of years of education (subjectively reported).
  years | 16.0 (3.2) | 15.7 (3.1) | 15.9 (3.2)
DHA Intake at Screening [Mean (Standard Deviation); unit: mg/day] — DHA Food Frequency Scale Total - a one page questionnaire asking about total monthly dietary intake of items such as fish, shellfish, turkey, chicken, beef, egg yolks, and liver.
  mg/day | 119.9 (77.4) | 148.7 (88.1) | 134.8 (82.9)
MoCA Score [Mean (Standard Deviation); unit: units on a scale] — The MoCA is a short cognitive screening test designed to assist health care professionals for the detection of mild cognitive impairment. The MoCA is scored on a 0 to 30 scale, with lower numbers indicating more cognitive impairment. A point is added to the MoCA if the subject's education high school or less (12 years or less education). Scores ranging from 26 - 30 are normal, 18 - 26 mild impairment, 10 - 17 moderate impairment, and less than 10 severe cognitive impairment.
  units on a scale | 25.1 (3.8) | 24.7 (2.6) | 24.9 (3.2)
Unified Parkinsons Disease Rating Scale (UPDRS-III) [Mean (Standard Deviation); unit: units on a scale] — This is the motor subsection of the Unified Parkinson's Disease Rating Scale (UPDRS) and is a commonly used tool to rate the symptoms of Parkinson's disease. Each item on the scale is rated from 0 (normal) to 4 (Can barely perform the task) several motor areas including speech, facial expression, tremor, rigidity, hand movements, agility, posture, and gait. Total score ranges from 0 to 108 with higher values on this scale represent a more severe stage of the disease.
  units on a scale | 34.6 (9.7) | 29.2 (10.9) | 31.9 (10.5)
Hoehn & Yahr [Median (Full Range); unit: units on a scale] — This is an objective staging scale for rating the clinical functioning of Parkinson's disease patients, combining functional deficits (disability) and objective signs (impairment). This staging scale is commonly used in both research settings and clinical practice. The Hoehn & Yahr is an ordinal scale ranging from 0 (no signs of disease) to 5 (wheelchair bound/bedridden). The modified version of the scale includes increments of 0.5. The HY has shown good inter-rater reliability and, although it is used worldwide, the clinimetric validity has not been established.
  units on a scale | 2.5 [2.0 to 3.0] | 2.0 [2.0 to 3.0] | 2.25 [2.0 to 3.0]
Levodopa Initial Dose [Median (Full Range); unit: mg/day] — Initial dose of levodopa (carbidopa/levodopa or Sinemet) as prescribed by treating physician in mg/day. This oral levodopa dose was prescribed clinically and is the first prescription of Sinemet (carbidopa/levodopa) that the participant ever received.
  mg/day | 300.0 [150 to 400] | 300.0 [300 to 600] | 300.0 [150 to 600]
Levodopa Exposure (Equivalence) [Median (Full Range); unit: mg/day] — Prior levodopa exposure as measured by subjective self report and medical record review for dopamine agonists (such as amantadine, apomorphine, pramipexole, ropinirole, rotigotine). Converted to levodopa equivalence using the Parkinson's UK Levodopa Equivalent Dose Calculator. This is levodopa exposure prior to starting Sinemet (carbidopa/levodopa), prior to entry into the study, through another drug like a dopamine agonist.
  mg/day | 540.0 [330.0 to 1440.0] | 187.5 [30.0 to 1425.0] | 345.0 [30.0 to 1425.0]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of DHA - Change in Blood ng/dL Levels
Description: Therapeutic level monitoring will be accomplished by analyzing blood levels for DHA.
Time Frame: baseline and 1.5 years
Measure: Mean (Standard Deviation); unit: ng/dL - Blood
Arm/Group | Docosahexaenoic Acid | Placebo:
Number analyzed (Participants) | 13 | 15
ng/dL - Blood | 102.18 (50.0) | -13.20 (33.12)

2. Primary Outcome: Efficacy of DHA - Number of Participants With An Abnormal Safety Lab (CBC)
Description: This study is seeking to determine the safety/efficacy of DHA in Parkinson's disease patients. The safety/efficacy of DHA will be determined using periodic safety lab information. Safety labs for complete blood count (CBC) were performed at each inpatient visit, reviewed by the PI, and marked as normal or abnormal.
Time Frame: Year 1
Population: 3 participants did not complete year 1 visit (2 withdrew prior to year 1, 1 refused to travel for visit), 2 blood samples were hemolyzed and could not be analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Docosahexaenoic Acid | Placebo:
Number analyzed (Participants) | 11 | 14
Participants | 0 | 0

3. Secondary Outcome: Forceplate Measured Dyskinesia
Description: Dyskinesia are abnormal movements caused by levodopa. These abnormal movements will be measured with a forceplate (a device that is similar to a door mat). Dyskinesia will be examined at all inpatient visits and area under the curves will be compared with a clinical rating scale to measure the development of dyskinesia after starting levodopa therapy.
Time Frame: baseline and 1.5 years
Population: Docosahexaenoic Acid Arm: 2 participants withdrew after the 6 week visit, 4 didn't complete visit 5 due to: wife's death, too busy, new diagnosis of cancer.
Measure: Count of Participants; unit: Participants
Arm/Group | Docosahexaenoic Acid | Placebo:
Number analyzed (Participants) | 9 | 15
Participants
  Dyskinesia Present | 3 | 6
  Dyskinesia Absent | 6 | 9

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected over 1.5 years. Regular monthly phone calls were placed to participants to ask about adverse events, hospitalizations, and changes in medications. Adverse events were also gathered at the in-person visit occurring at 0 weeks, 6 weeks, 24 weeks, 52 weeks, and 72 weeks.
Arm/Group | Docosahexaenoic Acid | Placebo:
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/15
Other Adverse Events (participants affected / at risk) | 6/15 | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docosahexaenoic Acid (N=15) | Placebo: (N=15)
Prostate Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) — New diagnosis of prostate cancer.
Syncope (Nervous system disorders) | 0 (0) | 1 (1) — Syncope during IV infusion leading to discontinuing infusion, ER visit with overnight Hospitalization with no findings.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docosahexaenoic Acid (N=15) | Placebo: (N=15)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Urinary Track Infection (Infections and infestations) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes